CLINICAL TRIAL: NCT05468255
Title: The Impact of Removal of Exercise on Glycemic Control and Vascular Health in Older Active
Brief Title: The Impact of Removal of Exercise on Glycemic Control and Vascular Health in Older Active Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Leryn Reynolds, Assistant Professor, Old Dominion University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AGEGLYFMD
Record Dates: First submitted 2022-05-09; First posted 2022-07-21 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Glucose Intolerance; Exercise; Vascular Function
MeSH Terms: conditions — Glucose Intolerance; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Metabolic (Experimental): Metabolic: Participants will have their blood glucose levels measured via continuous glucose monitoring for 3 days while participating in their normal exercise routines (EX). Participants will also have their blood glucose levels measured for 3 days while not exercising (NOEX), following immediately by 3 days of a return to normal activity(REX). Participants will be randomized to participate in the EX or NOEX/REX phases first. The EX and NOEX/REX phases will be separated by at least 1 week
  Interventions: Other: removal of exercise
- Vascular (Experimental): Vascular: Participants will have their blood vessel health measured while performing their normal exercise routines (EX) and while undergoing 1, 3, 5 days of no exercise (NOEX) followed immediately by 1 and 3 days of return to exercise (REX).
  Interventions: Other: removal of exercise

INTERVENTIONS:
Other: removal of exercise — Subjects will stop doing their normal exercise routines for 3 or 5 days and then subjects will resume doing their normal exercise routines for 3 days.
  Other Names: return to exercise

SUMMARY:
The purpose of this study is to determine if an acute bout of removal of exercise reduces enothelial function and glycemic control in an active, older adult population; and whether a 3 day return to exercise restores this response. Glycemic control is the blood glucose response following the consumption of a meal. It is an indicator of insulin resistance (or type 2 diabetes) and impaired glycemic control has been suggested to lead to cardiovascular disease. Endothelial function has been shown to be improved by chronic or acute increases in physical activity. Both of these have been shown to be impaired to acute bouts of inactivity in young populations; however the impact of acute inactivity in older adults is less understood. In this proposal the investigators will examine 1)how quickly impairments in glycemic control occur to acute physical inactivity in older adults who exercise, 2) how quickly impairments in endothelial function occur to acute inactivity in older adults who exercise, and 3) whether 3 days of a return to exercise restores these responses.

ELIGIBILITY:
Inclusion Criteria:

1. 55 years and older, 18-40 years old
2. Healthy, physically active, performing at least 90 min/week of physical activity
3. Free of physical limitations that may interfere with alterations in daily physical activity levels

Exclusion Criteria:

1. Physician diagnosed HIV, hepatitis, or tuberculosis.
2. Body weight change of greater than 5% within the previous 2 months
3. Smoking within the previous 2 months.
4. Taking medications that alter blood glucose levels

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Continuous glucose monitoring | 3 days before removal of exercise
Continuous glucose monitoring | After removal of exercise for 5 days
Continuous glucose monitoring | After return to exercise for 3 days
Flow mediated dilation | 3 days before removal of exercise
  This measure assess blood vessel health non-invasively
Flow mediated dilation (vascular health) | After removal of exercise for 5 days
  This measure assess blood vessel health non-invasively
Flow mediated dilation (vascular health) | After return to exercise for 3 days
  This measure assess blood vessel health non-invasively

CONTACTS AND LOCATIONS:
Locations (1):
- Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided